CLINICAL TRIAL: NCT00590317
Title: Ondansetron vs Prochlorperazine for Nausea and Vomiting in the Emergency Department
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Daniel Wu, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0998-2005
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Prochlorperazine; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prochlorperazine (Active Comparator): Patients receiving Prochlorperazine 10mg IV
  Interventions: Drug: Prochlorperazine
- Ondansetron (Active Comparator): Patient receiving Ondansetron 4mg IV
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Prochlorperazine — Patients receiving Prochlorperazine
  Arms: Prochlorperazine
Drug: Ondansetron — Patients receiving Ondansetron
  Arms: Ondansetron

SUMMARY:
This study will compare the effect of prochlorperazine and ondansetron for the treatment of nausea and vomiting in the emergency department.

DETAILED DESCRIPTION:
Nausea and vomiting can be common symptoms in the emergency department (ED). Antiemetics, agents to treat nausea and vomiting, include phenothiazine derivatives, prokinetic agents, and 5-HT3 antagonists. There have been limited studies on the use of these agents in the ED, and no direct comparisons to 5-HT3 antagonists have been published to date.

Inclusion Criteria:

Patients presenting to the ED with at least one of the following

* nausea
* vomiting documented in the ED

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the ED with at least one of the following
* Nausea
* Vomiting documented in the ED

Exclusion Criteria:

* Previous treatment in the ED with Ondansetron, prochlorperazine, promethazine or metaclopramide
* Patients with missed last menstrual period
* Pregnancy
* Age < 18 years old
* Treatment with antineoplastic agents within 7 days prior to randomization
* Irritable bowel syndrome
* Gastroparesis
* Suspected gastrointestinal bleed
* Suspected intestinal obstruction
* Preexisting motor disorder (Restless-leg syndrome or Parkinson's disease)
* Traumatic brain injury upon admission to ED
* Intracranial hemorrhage upon admission to ED
* Patients unable to read, write or communicate in the English language
* Patients leaving the ED against medical advice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Patka, PharmD, Principal Investigator — Grady Memorial Hospital; Daniel T Wu, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Hospital, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at one site (Hospital Emergency Department)over a period of March 2005 to September 2008
Pre-assignment Details: Patients were excluded if they chose to not participate after being enrolled and receiving medication but did not want to wait be observed for the 120 minute evaluation period.
Groups:
- Prochlorperazine: Patients receiving Prochlorperazine 10 mg IV
- Ondansetron: Patients receiving Ondansetron 4mg IV
Period: Overall Study
Arm/Group | Prochlorperazine | Ondansetron
Started | 32 | 32
Completed | 31 | 27
Not Completed | 1 | 5
Not completed — Lack of Efficacy | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Ondansetron: Patients receiving Ondansetron 4 mg IV
- Total: Total of all reporting groups
Arm/Group | Prochlorperazine | Ondansetron | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12) | 40 (11) | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Vomiting at 0 to 120 Min.
Time Frame: 0 to 120 minutes after receiving medication
Population: Convenience sample
Measure: Number; unit: number of participants exp vomiting
Arm/Group | Prochlorperazine | Ondansetron
Number analyzed (Participants) | 32 | 32
number of participants exp vomiting | 1 | 4

2. Secondary Outcome: Nausea at 0 to 120 Min
Description: 100mm Visual Analog scale (VAS) Scale is from 0 mm to 100 mm 0mm = no nausea 100mm = severe nausea
Time Frame: 0 to 120 minutes after receiving medication
Measure: Geometric Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prochlorperazine | Ondansetron
Number analyzed (Participants) | 32 | 32
units on a scale | 16.8 (21.9) | 34.3 (31.7)

3. Secondary Outcome: Akithisia at 0 to 120 Min
Time Frame: 0 to 120 min after receiving medication
Measure: Number; unit: no. participants exp akathisia
Arm/Group | Prochlorperazine | Ondansetron
Number analyzed (Participants) | 32 | 32
no. participants exp akathisia | 3 | 1

ADVERSE EVENTS:
Arm/Group | Prochlorperazine | Ondansetron
Serious Adverse Events (participants affected / at risk) | 3/32 | 1/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prochlorperazine (N=32) | Ondansetron (N=32)
Akathisia (Nervous system disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size due to limited enrollment. Fewer patient in the Odansetron group were discharged home suggesting a possibly sicker baseline group. Complete data sets were not available for all patients due to sedation and participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No